CLINICAL TRIAL: NCT03232138
Title: Randomized Clinical Trial of Lung Cancer Chemoprevention With Sulforaphane in Former Smokers
Brief Title: Clinical Trial of Lung Cancer Chemoprevention With Sulforaphane in Former Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jian-Min Yuan, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jian-Min Yuan, MD, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY19040278; R01CA213123 (NIH)
Record Dates: First submitted 2017-07-21; First posted 2017-07-27 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
Keywords: Sulforaphane; Chemoprevention; Former Smokers
MeSH Terms: conditions — Lung Neoplasms; Smoking Cessation | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulforaphane (Study Drug) (Experimental): Sulforaphane four tablets 2 times per day with breakfast and dinner each dose contains approximately 120 micromole of Sulforaphane
  Interventions: Dietary Supplement: Sulforaphane
- Placebo (Placebo Comparator): Placebo (containing no active drug) four tablets 2 times per day with breakfast and dinner
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Sulforaphane — Sulforaphane (SF) is a naturally occurring substance (phytochemical) found in cruciferous vegetables.
  Other Names: Avmacol®
  Arms: Sulforaphane (Study Drug)
Drug: Placebo — Inactive ingredients
  Arms: Placebo

SUMMARY:
This research study involves taking an experimental anti-cancer dietary supplement called Sulforaphane (SF) or a placebo (product without any supplement content) over a period of twelve months in order to determine if it is a useful dietary supplement for prevention of lung cancer in humans.

The main goals of this research study are:

1. To learn about the effects of giving Sulforaphane (SF) to former smokers who are still at high risk of developing cancer due to their smoking history and whether or not their condition improves, stays the same or becomes worse after Sulforaphane (SF) is given.
2. To learn whether Sulforaphane (SF) might reverse some of the lung cell changes associated with future development of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman 55-75 years of age.
2. Patients with normal endobronchial biopsy findings or pre-cancerous lesions at baseline will be eligible for the study. Pre-cancerous lesions include (a) reserve cell hyperplasia, (b) squamous metaplasia, (c) mild dysplasia, (d) moderate dysplasia, and (e) severe dysplasia.
3. A former smoker who has a history of smoking with ≥30 pack-years, quits smoking within the past 10 years, and has ≥1 year sustained abstinence from smoking.
4. Female subjects must be of non-child bearing potential or must have a negative serum pregnancy test at screening (within 72 hours of first dose of study medication) if of childbearing potential.
5. Male and female subjects of childbearing potential must be willing to use adequate barrier methods of contraception from the time starting with the screening visit through 30 days after the last dose of study therapy.
6. Abstinence is acceptable if this is the established and preferred contraception for the subject.
7. Generally healthy with liver enzyme and blood count values within the ranges shown below on the blood sample drawn at the baseline screening visit. Specifically:

   White blood cells ≥ 3,000/mL Total bilirubin ≤ 1.5 x ULN (upper limits of normal) AST (SGOT)/ALT (SGPT) ≤ 2.5 x ULN BUN and serum creatinine ≤ 1.5 x ULN Serum pregnancy test Negative
8. The presence of airflow obstruction on spirometry (GOLD II or greater, Forced Expiratory Volume in the first second (FEV1) <80%) Chronic Obstructive Pulmonary Disease (COPD); and/or any emphysema on CT scan.
9. Participants must have a Southwest Oncology Group (SWOG) performance status of 0-2
10. Participants must be able and willing to undergo a bronchoscopy before and after treatment for 12 months.
11. Patients must be fully informed of the investigational nature of this study and must sign an informed consent in accordance within institutional and regulatory guidelines.

Exclusion Criteria:

1. Carcinoma in situ or invasive cancer on baseline endobronchial biopsy.
2. A malignancy except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
3. Severe lung disease or inability to undergo two bronchoscopies.
4. Had pneumonia or acute bronchitis for at least 2 weeks prior to enrollment.
5. Cardiac dysrhythmia that is potentially life-threatening, such as ventricular tachycardia, multifocal premature ventricular contractions or supraventricular tachycardias with a rapid ventricular response. Well-controlled atrial fibrillation or rare (< 2 minutes) premature ventricular contractions are not exclusionary.
6. Evidence of clinically active coronary artery disease, including myocardial infarction within 6 weeks, chest pain, or congestive heart failure, or any serious medical condition which would preclude a patient from undergoing a bronchoscopy or would jeopardize the goals of the study.
7. Hypoxemia (less than 90% saturation with supplemental oxygen).
8. Prior chemotherapy or thoracic radiation within the past 5 years.
9. Woman who is pregnant or plan to be pregnant in next 12 months, or is breast feeding or plan to begin breast feeding in next 12 months.
10. Life expectancy of < 12 months.
11. Have a history of irritable bowel disease such as Crohn's disease and ulcerative colitis.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Min Yuan, MD, PhD, Principal Investigator — Univesity of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sulforaphane (Study Drug) | Placebo
Started | 21 | 22
Completed | 17 | 20
Not Completed | 4 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: We conducted telephone screening interview for eligibility on 105 subjects, of whom 67 were potentially eligible for the study. Of the 67 who visited our research clinic, 47 passed the physical examination and clinical tests. We randomized 43 participants after 4 eligible subjects declined to participate in the study. Of those randomized, 37 (17 in the SFN arm and 20 in the placebo arm) completed the entire course of the study and 7 (5 in the SFN arm and 2 in the placebo arm) withdrew.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulforaphane (Study Drug) | Placebo | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (5.3) | 68.0 (3.2) | 66.2 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 20 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 19 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education levels [Count of Participants; unit: Participants]
  High school or less | 3 | 5 | 8
  College | 12 | 11 | 23
  Graduate school | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bronchial Dysplasia Index at 12 Months
Description: To explore if daily oral dose of 120 micromole SF can modulate the changes in bronchial dysplasia from endoscopic biopsies in former smokers at high risk for lung cancer. All bronchial biopsies were formalin fixed, paraffin embedded, and H&E stained for subsequent morphologic evaluation and classification defined by the World Health Organization The scale to score the biopsy: 1= normal; 2= reserve cell hyperplasia; 3 = squamous metaplasia; 4 = mild dysplasia; 5 = moderate dysplasia; 6 = severe dysplasia; 7 = carcinoma in situ; and 8 = invasive carcinoma. The higher the score the worse the possible outcome.
Time Frame: 12 months
Population: Mean change from pre to post treatment (95%) confidence interval.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Sulforaphane (Study Drug) | Placebo
Number analyzed (Participants) | 17 | 20
score
  Pre treatment | 1.67 (0.38) | 1.62 (0.41)
  Post treatment | 1.55 (0.44) | 1.48 (0.37)
Statistical Analysis 1: Comparison: Sulforaphane (Study Drug); Derived from ANCOVA model with adjustment for baseline average endobronchial histopathological scores, age, sex, cigarettes per day, years of smoking, and years since quit smoking; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.452, ANCOVA — Hypothesis: sulforaphane treatment slows or reverse the progression of lung histological lesions or lower the dysplasia score; ANCOVA model includes baseline average endobronchial histopathological scores,age,sex,cigarettes per day,years of smoking, years since quit smoking; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [0.03 to 0.41]
Statistical Analysis 2: Comparison: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.452, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.04 to 0.28]

2. Primary Outcome: Cell Proliferation Marker Ki-67
Description: The primary outcome focuses on the changes of bronchial dysplasia index with cell proliferation marker Ki-67. The determination if a daily oral dose of 120 micromole SF for 12 months can modulate the changes of bronchial dysplasia index, cell proliferation marker Ki-67. Besides the inhibition of tumor incidence and multiplicity, the use of sulforaphane can inhibit cellular proliferation markers such as Ki-67 and induction of apoptosis hallmarks of tumorigenesis. Ki-67 will be quantified as % positive cells in two slides of each tissue block. First, we calculate the average values of each of the 3 IHC markers over 6 tissue blocks within each bronchoscopy per patient separately for pre- and post-treatment. The primary analysis for these continuous measures will be a linear regression predicting post-treatment score by treatment group, controlling for pre-treatment score.
Time Frame: 12 months
Population: Mean changes from the baseline and pre to post treatment.
Measure: Mean (95% Confidence Interval); unit: counts per µm^2
Arm/Group | Sulforaphane (Study Drug) | Placebo
Number analyzed (Participants) | 17 | 20
counts per µm^2
  Baseline: All positive nuclei | 26.07 [18.64 to 33.51] | 27.75 [24.90 to 34.61]
  Baseline: Weak-Intensity positive nuclei | 11.71 [8.85 to 14.57] | 12.21 [9.57 to 14.85]
  Baseline: Moderate Intensity positive nuclei | 6.70 [4.42 to 8.97] | 7.22 [5.12 to 9.32]
  Baseline: Strong intensity positive nuclei | 7.67 [4.61 to 10.72] | 8.32 [5.51 to 11.14]
  Pre to Post Treatment: All positive nuclei | -5.27 [-18.13 to 7.59] | 18.03 [7.18 to 28.88]
  Pre to Post Treatment: Weak-intensity positive nuclei | -0.50 [-6.44 to 5.26] | 7.48 [2.55 to 12.41]
  Pre to Post Treatment: Moderate-intensity positive nuclei | -1.16 [-4.76 to 2.44] | 4.61 [1.57 to 7.64]
  Pre to Post Treatment: Strong-intensity positive nuclei | -3.41 [-7.67 to 0.85] | 5.93 [2.24 to 9.52]
Statistical Analysis 1: Comparison: Sulforaphane (Study Drug) vs Placebo; All positive nuclei. Mean (95%CI) changes in baseline; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.738, Analysis of Covariance — Hypothesis: Sulforaphane treatment inhibits or reduces number of Ki-67 positive nuclei in bronchial biopsy as compared with the placebo
Statistical Analysis 2: Comparison: Sulforaphane (Study Drug) vs Placebo; Weak-intensity positive nuclei. Mean (95%CI) baseline; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.780, Analysis of Covariance — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Sulforaphane (Study Drug) vs Placebo; Moderate intensity positive nuclei. Mean (95%CI) changes in baseline; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.733, Analysis of Covariance — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Sulforaphane (Study Drug) vs Placebo; Strong-Intensity positive nuclei. Mean (95%CI) changes in baseline; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.751, Analysis of Covariance — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Sulforaphane (Study Drug) vs Placebo; All positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.014, Analysis of Covariance — [p-value comment as in outcome 2, analysis 1]; Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking, baseline values of Ki-67 positive nuclei
Statistical Analysis 6: Comparison: Sulforaphane (Study Drug) vs Placebo; Week intensity positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.056, Covariance; Analysis of Covariance adjustment age, sex, cigarettes/day, years of smoking, years of quit smoking,baseline values of the same cellular biomarker
Statistical Analysis 7: Comparison: Sulforaphane (Study Drug) vs Placebo; Moderate Intensity positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.028, Analysis of Covariance; Analysis of Covariance adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking,baseline values of the same cellular biomarker
Statistical Analysis 8: Comparison: Sulforaphane (Study Drug) vs Placebo; Strong intensity positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.004, Analysis of Covariance; [statistical method as in outcome 2, analysis 7]

3. Primary Outcome: Apoptosis Marker TUNEL
Description: The determination if a daily oral dose of 120 micromole SF for 12 months can modulate the changes of bronchial dysplasia index, in apoptosis marker TUNEL in bronchial biopsies in former smokers at high risk for lung cancer. TUNEL will be quantified as % positive cells in two slides of each tissue block. First, we calculate the average values of each of the 3 IHC markers over 6 tissue blocks within each bronchoscopy per patient separately for pre- and post-treatment. The primary analysis for these continuous measures will be a linear regression predicting post-treatment score by treatment group, controlling for pre-treatment score.
Time Frame: 12 months
Population: TUNEL positive nuclei (counts/µm2) Mean (95% CI) changes from baseline and pre- to post-treatment
Measure: Mean (95% Confidence Interval); unit: counts/µm2
Arm/Group | Sulforaphane (Study Drug) | Placebo
Number analyzed (Participants) | 17 | 20
counts/µm2
  Baseline: All positive nuclei | 5.01 [4.28 to 5.75] | 4.57 [3.89 to 5.25]
  Baseline: Weak-intensity positive nuclei | 2.73 [2.33 to 3.13] | 2.51 [2.15 to 2.88]
  Baseline: Moderate-intensity positive nuclei | 1.78 [1.52 to 2.04] | 1.61 [1.37 to 1.85]
  Baseline: Strong-intensity positive nuclei | 0.50 [0.37 to 0.63] | 0.45 [0.33 to 0.57]
  Pre to Post Treatment: All positive nuclei | -0.21 [-0.96 to 0.53] | 0.35 [-0.27 to 0.96]
  Pre to Post Treatment: Weak-intensity positive nuclei | -0.05 [-0.43 to 0.34] | 0.12 [-0.27 to 0.44]
  Pre to Post Treatment: Moderate-intensity positive nuclei | -0.10 [-0.38 to 0.18] | 0.16 [-0.08 to 0.39]
  Pre to Post Treatment: Strong-intensity positive nuclei | -0.05 [-0.18 to 0.09] | 0.05 [-0.06 to 0.17]
Statistical Analysis 1: Comparison: Sulforaphane (Study Drug) vs Placebo; All positive nuclei. Mean (95%CI) baseline; Test type: Equivalence — 2-sided P-value in the analysis, Mean (95%CI) at baseline for positive cells. TUNEL positive nuclei (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarker; p = 0.377, Analysis of Covariance — Hypothesis: Sulforaphane treatment has significant impact on number of TUNEL positive nuclei in bronchial biopsies compared with the place; Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking, baseline values of positive TUNEL nuclei
Statistical Analysis 2: Comparison: Sulforaphane (Study Drug) vs Placebo; Weak-intensity positive nuclei. Mean (95%CI) baseline; Test type: Equivalence — 2-sided P-value in the analysis; p = 0.413, Analysis of Covariance — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Sulforaphane (Study Drug) vs Placebo; Moderate Intensity positive nuclei. Mean (95%CI) at baseline; Test type: Equivalence — 2-sided P-value in the analysis, Mean (95%CI) at baseline Moderate-intensity positive nuclei. TUNEL positive (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarker; p = 0.338, Analysis of Covariance — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Sulforaphane (Study Drug) vs Placebo; Strong-intensity positive nuclei. Mean (95%CI) baseline; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.547, Analysis of Covariance — Hypothesis: Sulforaphane treatment has significant impact on number of TUNEL positive nuclei in bronchial biopsies; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Sulforaphane (Study Drug) vs Placebo; All positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — used 2-sided P-value in the analysis, Mean (95%CI) changes from pre to pos treatment for all positive cells. TUNEL all positive nuclei (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarker; p = 0.291, Analysis of Covariance — Hypothesis: Sulforaphane treatment has significant impact on number of TUNEL positive nuclei in bronchial biopsies; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Sulforaphane (Study Drug) vs Placebo; Weak-intensity positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — 2-sided P-value in the analysis, Mean (95%CI) changes from pre to pos treatment for positive cells. TUNEL all positive nuclei (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarker; p = 0.552, Analysis of Covariance — Hypothesis: Sulforaphane treatment has significant impact on number of TUNEL positive nuclei in bronchial biopsies; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Sulforaphane (Study Drug) vs Placebo; Moderate-intensity positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — [test comment as in outcome 3, analysis 6]; p = 0.205, Analysis of Covariance — Hypothesis: Sulforaphane treatment has significant impact on number of TUNEL positive nuclei in bronchial biopsies; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Sulforaphane (Study Drug) vs Placebo; Strong-intensity positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — [test comment as in outcome 3, analysis 6]; p = 0.295, Analysis of Covariance — Hypothesis: Sulforaphane treatment has significant impact on number of TUNEL positive nuclei in bronchial biopsies; [statistical method as in outcome 3, analysis 1]

4. Primary Outcome: Apoptosis Marker Caspase-3
Description: The determination if a daily oral dose of 120 micromole SF for 12 months can modulate the changes of bronchial dysplasia index, in apoptosis marker Caspase-3 in bronchial biopsies in former smokers at high risk for lung cancer. Caspase-3 will be quantified as % positive cells in two slides of each tissue block. First, we calculate the average values of each of the 3 IHC markers over 6 tissue blocks within each bronchoscopy per patient separately for pre- and post-treatment. The primary analysis for these continuous measures will be a linear regression predicting post-treatment score by treatment group, controlling for pre-treatment score.
Time Frame: 12 months
Population: Caspase-3 positive cytoplasm (% of total cells examined)
Measure: Mean (95% Confidence Interval); unit: percent of cells
Arm/Group | Sulforaphane (Study Drug) | Placebo
Number analyzed (Participants) | 17 | 20
percent of cells
  Baseline: All positive cells | 4.46 [2.36 to 6.57] | 2.96 [1.02 to 4.90]
  Baseline: Weak-intensity positive cells | 4.18 [2.31 to 6.04] | 2.69 [0.97 to 4.41]
  Baseline: Moderate-intensity positive cells | 0.25 [-0.01 to 0.50] | 0.25 [0.01 to 0.49]
  Baseline: Strong-intensity positive cells | 0.04 [-0.002 to 0.08] | 0.02 [-0.02 to 0.06]
  Pre to Post Treatment: All positive cells | -1.28 [-2.64 to 0.08] | -1.00 [-2.15 to 0.96]
  Pre to Post Treatment: Weak-intensity positive cells | -1.19 [-2.44 to 0.06] | -0.83 [-1.88 to 0.23]
  Pre to Post Treatment: Moderate-intensity positive cells | -0.07 [-0.21 to 0.08] | -0.14 [-0.26 to -0.02]
  Pre to Post Treatment: Strong-intensity positive cells | -0.01 [-0.02 to -0.001] | -0.03 [-0.04 to -0.02]
Statistical Analysis 1: Comparison: Sulforaphane (Study Drug) vs Placebo; All positive nuclei. Mean (95%CI) at baseline; Test type: Equivalence — 2-sided P-value in the analysis, Mean (95%CI) baseline positive cells. Caspase-3 positive nuclei (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarker; p = 0.295, Analysis of Covariance — Hypothesis: Sulforaphane treatment has significant impact on the number of cells with positive Caspase-3 in bronchial biopsies than the placebo; Analysis of Covariance adjustment for age,sex,cigarettes/day,years of smoking,years of quit smoking,baseline values of Caspase-3 positive cells
Statistical Analysis 2: Comparison: Sulforaphane (Study Drug) vs Placebo; weak intensity positive nuclei. Mean (95%CI) at baseline; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.242, Analysis of Covariance — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Sulforaphane (Study Drug) vs Placebo; Moderate intensity positive nuclei. Mean (95%CI) at baseline; Test type: Equivalence — -sided P-value in the analysis, Mean (95%CI) baseline positive cells. Caspase-3 positive nuclei (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarker; p = 0.985, Analysis of Covariance — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Sulforaphane (Study Drug) vs Placebo; Strong intensity positive nuclei. Mean (95%CI) at baseline; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.547, Analysis of Covariance — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Sulforaphane (Study Drug) vs Placebo; All positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — used 2-sided P-value in the analysis, Mean (95%CI) changes from pre to pos treatment for all positive cells. Caspase-3 all positive nuclei (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarker; p = 0.778, Analysis of Covariance — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Sulforaphane (Study Drug) vs Placebo; Weak intensity positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — 2-sided P-value in the analysis, Mean (95%CI) changes from pre to pos treatment for positive cells. Caspase-3 all positive nuclei (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarker; p = 0.685, Analysis of Covariance — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Sulforaphane (Study Drug) vs Placebo; Moderate intensity positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — -sided P-value in the analysis, Mean (95%CI) changes from pre to pos treatment for positive cells. Caspase-3 all positive nuclei (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarker; p = 0.469, Analysis of Covariance — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Sulforaphane (Study Drug) vs Placebo; strong intensity positive nuclei. Mean (95%CI) changes from pre to pos treatment; Test type: Equivalence — 2-sided P-value in the analysis, Mean (95%CI) changes from pre to pos treatment for positive cells. Caspase-3 all positive nuclei (counts/µm2) From Analysis of Covariance with adjustment for age, sex, cigarettes/day, years of smoking, years of quit smoking and baseline values of the same cellular biomarke; p = 0.052, Analysis of Covariance — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Upregulated Genes Associated With Lung Cancer Risk in Bronchial Brushing Samples
Description: Gene set variation analysis (GSVA) algorithm was used to calculate gene set enrichment scores in bronchial brushing samples. If a gene is upregulated in lung cancer (LC) tissue, the inhibitory effect of sulforaphane (SFN) treatment on such genes suggests a protective effect against LC.
Time Frame: 12 Months
Population: Due to poor quality of RNA and missing data on the gene expression, we excluded 5 subjects in the sulforaphane group and 4 subjects in the placebo group. The final analysis for this secondary outcome included 12 subjects in the sulforaphane and 16 subjects in the placebo group.
Measure: Mean (Standard Deviation); unit: Relative score from -1 to +1
Units Other Than Participants: Upregulated genes with lung cancer risk
Groups:
- Sulforaphane: Sulforaphane four tablets 2 times per day with breakfast and dinner each dose contains approximately 120 micromole of Sulforaphane Sulforaphane: Sulforaphane (SF) is a naturally occurring substance (phytochemical) found in cruciferous vegetables.
- Placebo: Placebo (containing no active drug) four tablets 2 times per day with breakfast and dinner for 12 months.
  Placebo: Inactive ingredients
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 12 | 16
Number analyzed (Upregulated genes with lung cancer risk) | 44 | 44
Relative score from -1 to +1
  Gene enrichment score pre-treatment | 0.04 (0.25) | 0.02 (0.26)
  Gene enrichment score post-treatment | 0.03 (0.32) | -0.02 (0.31)
Statistical Analysis 1: Comparison: Sulforaphane; Test type: Equivalence — This analysis was focused on the gene set that were found to be upregulated in lung cancer. the objective was to examine if sulforaphane treatment for 12 months had any significant impact on the expression of these lung-cancer associated upregulated genes in bronchial brushing samples. A linear mixed model was used to evaluate the effect of sulforaphane treatment over time on GSVA enrichment score with adjustment for age at study entry, sex, and RNA integrity number or RIN; p = 0.82, Mixed Models Analysis — Hypothesis: Sulforaphane treatment downregulate these genes whose over-expressions are associated with risk of lung cancer; The model includes treatment, time, time*treatment, age at study entry, sex, and RIN; Slope = 0.02, Standard Error of Mean 0.10 — Changes (beta) of gene expression after 12-month sulforaphane treatment

6. Secondary Outcome: Downregulated Genes Associated With Lung Cancer Risk in Bronchial Brushing Samples
Description: Gene set variation analysis (GSVA) algorithm was used to calculate gene set enrichment scores in bronchial brushing samples. If a gene is downregulated in LC, the enhancing effect of sulforaphane (SFN) treatment on such genes suggests a protective effect against LC.
Time Frame: 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Relative score from -1 to +1
Units Other Than Participants: upregulated gene with lung cancer risk
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 12 | 16
Number analyzed (upregulated gene with lung cancer risk) | 113 | 113
Relative score from -1 to +1
  gene enrichment score pre-treatment | -0.10 (0.27) | -0.07 (0.25)
  gene enrichment score post-treatment | -0.03 (0.35) | 0.08 (0.28)
Statistical Analysis 1: Comparison: Sulforaphane vs Placebo; Test type: Equivalence — This analysis was focused on the gene set that were found to be down-regulated in lung cancer. The objective was to examine if sulforaphane treatment for 12 months had any significant impact on the expression of these lung-cancer associated down-regulated genes in bronchial brushing samples. A linear mixed model was used to evaluate the effect of sulforaphane treatment over time on GSVA enrichment score with adjustment for age at study entry, sex, and RIN; p = 0.50, Mixed Models Analysis — Hypothesis: Sulforaphane treatment would upregulate these genes whose down-expressions are associated with lung cancer risk; The model includes treatment, time, time*treatment, age at study entry, sex, and RIN; Slope = -0.07, Standard Error of Mean 0.10 — Changes (beta) of gene expression after 12-month sulforaphane treatment

7. Secondary Outcome: Upregulated Genes Associated With Lung Pre-Malignant Lesions (PML) in Bronchial Brushing Samples
Description: GSVA algorithm was used to calculate gene set enrichment scores in bronchial brushing samples. If a gene is upregulated in lung pre-malignant lesions (PML), the inhibitory effect of sulforaphane (SFN) treatment on such genes suggests a protective effect against PML.
Time Frame: 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: relative score from -1 to +1
Units Other Than Participants: Upregulated genes with PML risk
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 12 | 16
Number analyzed (Upregulated genes with PML risk) | 61 | 61
relative score from -1 to +1
  Upregulated gene enrichment score at pre-treatment | -0.27 (0.41) | -0.12 (0.46)
  Upregulated gene enrichment score at post-treatment | 0.15 (0.42) | 0.11 (0.41)
Statistical Analysis 1: Comparison: Sulforaphane vs Placebo; Test type: Equivalence — This analysis was focused on the gene set that were found to be upregulated in lung pre-malignant lesions. The objective was to examine if sulforaphane treatment for 12 months would have any significant impact on the expression of these pre-malignant lesions associated upregulated genes in bronchial brushing samples. A linear mixed model was used to evaluate the effect of sulforaphane treatment over time on GSVA enrichment score with adjustment for age at study entry, sex, and RIN; p = 0.32, Mixed Models Analysis — Hypothesis: Sulforaphane treatment would downregulate these genes whose over-expressions are associated with risk of lung pre-malignant lesions; The model includes treatment, time, time*treatment, age at study entry, sex, and RIN; Slope = 0.15, Standard Error of Mean 0.15 — Changes (beta) of gene expression after the 12-month sulforaphane treatment

8. Secondary Outcome: Downregulated Genes Associated With Lung Pre-malignant Lesions (PML) in Bronchial Brushing Samples
Description: GSVA algorithm was used to calculate gene set enrichment scores in bronchial brushing samples. If a gene is downregulated in PML, the enhancing effect of sulforaphane (SFN) treatment on such genes also suggests a protective effect against PML.
Time Frame: 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: relative score from -1 to +1
Units Other Than Participants: upregulated gene with PML cancer risk
Arm/Group | Sulforaphane (Study Drug) | Placebo
Number analyzed (Participants) | 12 | 16
Number analyzed (upregulated gene with PML cancer risk) | 153 | 153
relative score from -1 to +1
  Downregulated gene enrichment score at pre-treatment | 0.20 (0.37) | 0.11 (0.41)
  Downregulated gene enrichment score at post-treatment | -0.15 (0.40) | -0.12 (0.40)
Statistical Analysis 1: Comparison: Sulforaphane (Study Drug) vs Placebo; Test type: Equivalence — This analysis was focused on the gene set that were found to be downregulated in lung pre-malignant lesions. The objective was to examine if sulforaphane treatment for 12 months would have any significant impact on the expression of these pre-malignant lesions associated downregulated genes in bronchial brushing samples. A linear mixed model was used to evaluate the effect of sulforaphane treatment over time on GSVA enrichment score with adjustment for age at study entry, sex, and RIN; p = 0.5, Mixed Models Analysis — Hypothesis: Sulforaphane treatment would upregulate these genes whose down-regulated expressions are associated with risk of lung pre-malignant lesions; The model includes treatment, time, time*treatment, age at study entry, sex, and RIN; Slope = -0.10, Standard Error of Mean 0.14 — Changes (beta) of gene expression after the 12-month sulforaphane treatment

9. Secondary Outcome: Upregulated Genes Associated With Risk of Lung Cancer in Nasal Brushing Samples
Description: Similarly, GSVA algorithm was used to calculate gene set enrichment scores in nasal brushing samples. If a gene is upregulated in lung cancer (LC), the inhibitory effect of sulforaphane (SFN) treatment on such genes suggests a protective effect against LC.
Time Frame: 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: relative score from -1 to +1
Units Other Than Participants: Nasal upregulated genes with LC risk
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 12 | 16
Number analyzed (Nasal upregulated genes with LC risk) | 41 | 41
relative score from -1 to +1
  Gene enrichment score at pre-treatment | 0.22 (0.23) | 0.00 (0.29)
  Gene enrichment score at pre-treatment at post-treatment | -0.15 (0.17) | -0.07 (0.25)
Statistical Analysis 1: Comparison: Sulforaphane vs Placebo; Test type: Equivalence — This analysis was focused on the gene set that were found to be upregulated in lung cancer. The objective was to examine if sulforaphane treatment for 12 months had any significant impact on the expression of these lung-cancer associated upregulated genes in nasal brushing samples. A linear mixed model was used to evaluate the effect of sulforaphane treatment over time on GSVA enrichment score with adjustment for age at study entry, sex, and RIN; p = 0.012, Mixed Models Analysis — Sulforaphane treatment would downregulate the expression of these genes whose upregulated expressions in bronchial epithelial cells have been found to be associated with risk of lung cancer; The model includes treatment, time, time*treatment, age at study entry, sex, and RIN; Slope = -0.27, Standard Error of Mean 0.10 — Changes (beta) of gene expression after the 12-month sulforaphane treatment

10. Secondary Outcome: Downregulated Genes Associated With Risk of Lung Cancer in Nasal Brushing Samples
Description: GSVA algorithm was used to calculate gene set enrichment scores in nasal brushing samples. If a gene is downregulated in lung cancer (LC), the enhancing effect of sulforaphane (SFN) treatment on such genes also suggests a protective effect against LC.
Time Frame: 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: relative score from -1 to +1
Units Other Than Participants: Nasal upregulated genes with LC risk
Arm/Group | Sulforaphane (Study Drug) | Placebo
Number analyzed (Participants) | 12 | 16
Number analyzed (Nasal upregulated genes with LC risk) | 116 | 116
relative score from -1 to +1
  Gene enrichment score at pre-treatment | -0.29 (0.33) | 0.02 (0.37)
  Gene enrichment score at pre-treatment at post-treatment | 0.19 (0.32) | 0.06 (0.34)
Statistical Analysis 1: Comparison: Sulforaphane (Study Drug) vs Placebo; Test type: Equivalence — This analysis was focused on the gene set that were found to be downregulated in lung cancer. The objective was to examine if sulforaphane treatment for 12 months had any significant impact on the expression of these lung-cancer associated upregulated genes in nasal brushing samples. A linear mixed model was used to evaluate the effect of sulforaphane treatment over time on GSVA enrichment score with adjustment for age at study entry, sex, and RIN; p = 0.0045, Mixed Models Analysis — Hypothesis: Sulforaphane treatment would upregulate the expression of these genes whose downregulated expressions in nasal epithelial cells have been found to be associated with risk of lung cancer; Slope = 0.38, Standard Error of Mean 0.12 — Changes (beta) of gene expression after the 12-month sulforaphane treatment

11. Secondary Outcome: Upregulated Genes Associated With Risk of Lung Pre-malignant Lesions Cancer (PML) in Nasal Brushing Samples
Description: GSVA algorithm was used to calculate gene set enrichment scores in nasal brushing samples. If a gene is upregulated in PML. the inhibitory effect of sulforaphane (SFN) treatment on such genes suggests a protective effect against PML risk.
Time Frame: 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: relative score from -1 to +1
Units Other Than Participants: Nasal upregulated genes with LC risk
Arm/Group | Sulforaphane (Study Drug) | Placebo
Number analyzed (Participants) | 12 | 16
Number analyzed (Nasal upregulated genes with LC risk) | 60 | 60
relative score from -1 to +1
  Gene enrichment score at pre-treatment | -0.27 (0.42) | 0.08 (0.47)
  Gene enrichment score at pre-treatment at post-treatment | 0.08 (0.46) | 0.09 (0.46)
Statistical Analysis 1: Comparison: Sulforaphane (Study Drug) vs Placebo; Test type: Equivalence — This analysis was focused on the gene set that were found to be upregulated in lung premalignant lesions. The objective was to examine if sulforaphane treatment for 12 months had any significant impact on the expression of these premalignant lesion-associated upregulated genes in nasal brushing samples. A linear mixed model was used to evaluate the effect of sulforaphane treatment over time on GSVA enrichment score with adjustment for age at study entry, sex, and RIN; p = 0.32, Mixed Models Analysis — Hypothesis: Sulforaphane treatment would downregulate the expression of these genes whose upregulated expressions in bronchial epithelial cells have been found to be associated with risk of lung premalignant lesions; The model includes treatment, time, time*treatment, age at study entry, sex, and RIN; Slope = 0.17, Standard Error of Mean 0.16 — Changes (beta) of gene expression after the 12-month sulforaphane treatment

12. Secondary Outcome: Downregulated Genes Associated With Risk of Lung Pre-malignant Lesions (PML) in Nasal Brushing Samples
Description: Similarly, GSVA algorithm was used to calculate gene set enrichment scores in nasal brushing samples. If a gene is downregulated in PML, the overexpression effect of sulforaphane (SFN) treatment on such genes suggests a protective effect against PML
Time Frame: 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: relative score from -1 to +1
Units Other Than Participants: Nasal upregulated genes with LC risk
Arm/Group | Sulforaphane (Study Drug) | Placebo
Number analyzed (Participants) | 12 | 16
Number analyzed (Nasal upregulated genes with LC risk) | 155 | 155
relative score from -1 to +1
  Gene enrichment score at pre-treatment | 0.28 (0.38) | -0.12 (0.42)
  Gene enrichment score at pre-treatment at post-treatment | -0.01 (0.41) | -0.07 (0.42)
Statistical Analysis 1: Comparison: Sulforaphane (Study Drug) vs Placebo; Test type: Equivalence — This analysis was focused on the gene set that were found to be downregulated in lung premalignant lesions. The objective was to examine if sulforaphane treatment for 12 months had any significant impact on the expression of these premalignant lesion-associated downregulated genes in nasal brushing samples. A linear mixed model was used to evaluate the effect of sulforaphane treatment over time on GSVA enrichment score with adjustment for age at study entry, sex, and RIN; p = 0.27, Mixed Models Analysis — Hypothesis: Sulforaphane treatment would upregulate the expression of these genes whose downregulated expressions in bronchial epithelial cells have been found to be associated with risk of lung premalignant lesions; The model includes treatment, time, time*treatment, age at study entry, sex, and RIN; Slope = -0.16, Standard Error of Mean 0.14 — Changes (beta) of gene expression after the 12-month sulforaphane treatment

13. Secondary Outcome: Overall Number of Adverse Events That Occurred in the Study Population as Assessed by CTCAE v4.0
Description: To determine the safety and toxicity of daily oral dose of 120 micromole SF in former smokers at high risk for lung cancer by monitoring and recording any potential SF-related adverse events (both expected and unexpected events). The severity is calculated by five grades: 1=mild, 2 = moderate, 3 = severe, 4 = life threatening, 5 = death. Events are assigned to categories of unrelated, possibly elated, probably related, and related.
Time Frame: 12 Months
Population: Total number of adverse events by attrition and severity by treatment group during the study period, The Pittsburgh Clinical Trial of Sulforaphane (SFN) on Risk Markers of Lung Cancer. The number of patients included those who dropped out from the study.
Measure: Number; unit: events
Arm/Group | Sulforaphane (Study Drug) | Placebo
Number analyzed (Participants) | 21 | 22
events
  Unrelated Grade 1 | 56 | 66
  Unrelated Grade 2 | 17 | 12
  Unrelated Grade 3 | 1 | 3
  Unrelated Grade 4 | 0 | 0
  Unrelated Grade 5 | 0 | 0
  Possibly Related Grade 1 | 26 | 12
  Possibly Related Grade 2 | 3 | 5
  Possibly Related Grade 3 | 0 | 0
  Possibly Related Grade 4 | 0 | 0
  Possibly Related Grade 5 | 0 | 0
  Probably Related Grade 1 | 3 | 1
  Probably Related Grade 2 | 1 | 1
  Probably Related Grade 3 | 0 | 0
  Probably Related Grade 4 | 0 | 0
  Probably Related Grade 5 | 0 | 0
  Related Grade 1 | 0 | 0
  Related Grade 2 | 0 | 0
  Related Grade 3 | 0 | 0
  Related Grade 4 | 0 | 0
  Related Grade 5 | 0 | 0
  All adverse events Grade 1 | 85 | 79
  All adverse events Grade 2 | 21 | 18
  All adverse events Grade 3 | 1 | 3
  All adverse events Grade 4 | 0 | 0
  All adverse events Grade 5 | 0 | 0
Statistical Analysis 1: Comparison: Sulforaphane (Study Drug) vs Placebo; Test type: Equivalence — Total number of adverse events by attrition and severity by treatment group during the study period, The Pittsburgh Clinical Trial of Sulforaphane (SFN) on Risk Markers of Lung Cancer; p = 0.590, Fisher Exact — For severity by treatment group
Statistical Analysis 2: Comparison: Sulforaphane (Study Drug) vs Placebo; Test type: Equivalence — [test comment as in outcome 13, analysis 1]; p = 0.131, Fisher Exact — For attribution by treatment group

ADVERSE EVENTS:
Time Frame: 1 year treatment, 1year post treatment
Arm/Group | Sulforaphane (Study Drug) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 21/21 | 22/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulforaphane (Study Drug) (N=21) | Placebo (N=22)
Bad taste (Gastrointestinal disorders) | 1 | 3
Belching (Gastrointestinal disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 7 | 9
Diarrhea (Gastrointestinal disorders) | 10 | 9
Distension (Gastrointestinal disorders) | 3 | 3
Dry Mouth (Gastrointestinal disorders) | 6 | 9
Flatulence (Gastrointestinal disorders) | 13 | 13
Stomachache (Gastrointestinal disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 6 | 6
Vomiting (Gastrointestinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 6 | 7
Headache (Nervous system disorders) | 3 | 5
Mood Alteration (Nervous system disorders) | 7 | 7
Tremor (Nervous system disorders) | 5 | 1
Insomnia (General disorders) | 9 | 5
Others (General disorders) | 17 | 10

LIMITATIONS AND CAVEATS:
Limited study size due to the circumstances of COVID19 impact on in person research studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03232138/Prot_SAP_000.pdf